CLINICAL TRIAL: NCT04106076
Title: Phase I, Open Label Dose-escalation Study to Evaluate the Safety, Expansion, Persistence and Clinical Activity of Multiple Infusions of UCART123 (Allogeneic Engineered T-cells Expressing Anti-CD123 Chimeric Antigen Receptor) in Patients With Adverse Genetic Risk Acute Myeloid Leukaemia
Brief Title: Phase I Study of UCART123 in Patient With Adverse Genetic Risk Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was discontinued due to sponsor's decision and not a consequence of any safety concern
Sponsor: Cellectis S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCART123_03
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Acute Myeloid Leukaemia
Keywords: Acute Myeloid Leukaemia; Newly diagnosed AML; ELN adverse genetic risk group; Chimeric Antigen Receptor T-Cell (CAR-T) therapy; Allogeneic; Transcription Activator-Like Effector Nuclease (TALEN)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Several tested doses of UCART123 until the Maximum Tolerated Dose (MTD) is identified.
  Interventions: Biological: UCART123

INTERVENTIONS:
Biological: UCART123 — Allogeneic engineered T-cells expressing anti-CD123 Chimeric Antigen Receptor

SUMMARY:
This is a Phase I, open-label, dose escalation study of UCART123 administered intravenously to patients with newly diagnosed CD123 positive adverse genetic risk acute myeloid leukaemia (AML) defined in the ELN adverse genetic risk group (2017). The purpose of this study is to evaluate the safety and clinical activity of multiple infusions of UCART123 and to determine the Maximum Tolerated Dose (MTD).

ELIGIBILITY:
Main Inclusion Criteria:

* Patients newly diagnosed with CD123 positive adverse genetic risk acute myeloid leukaemia (AML) defined as per ELN guidelines (Döhner et al., 2017)
* Eastern Cooperative Oncology Group performance status of 0 or 1
* No prior gene or experimental cellular therapy
* No organ dysfunction that in the opinion of the investigator precludes intensive induction chemotherapy or cellular therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Incidence of AE/SAE/DLT [Safety and Tolerability] | 24 months
  Incidence, nature, and severity of adverse events and serious adverse events (SAEs) throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Mufti, Pr, Principal Investigator — Kings college London NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Undecided